CLINICAL TRIAL: NCT02756429
Title: Quantification of Endothelial Thrombogenicity in Patients With Atrial Fibrillation
Acronym: REMI-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2012-719
Record Dates: First submitted 2016-04-27; First posted 2016-04-29 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; stroke; thromboembolism; inflammation
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Thromboembolism; Inflammation | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- atrial fibrillation (Experimental): Patients with atrial fibrillation
  Interventions: Other: blood samples
- Control (Experimental): Patients without atrial fibrillation
  Interventions: Other: blood samples

INTERVENTIONS:
Other: blood samples — Patients with atrial fibrillation for whom electrophysiology exploration or ablation are programmed; All blood samples will be taken through the exploration catheter. For the peripheral blood sample, blood will be taken at the introduction of the catheter into the femoral vein. Then the blood samples in the coronary sinus and in the left atrium will be made at progressively exploration.

SUMMARY:
Atrial fibrillation (AF) is the most common cardiac arrhythmia. Because of its major impact on the general morbidity and risk of stroke, AF is a great concern for public health. Several mechanisms, including endothelial dysfunction and inflammatory processes, have been postulated as predisposing factors for AF, as well as for stroke.

Both clinical and experimental studies highlight inflammation as a predisposing factor for AF and its complications. Nevertheless, the source of high inflammatory proteins in patients with AF is still unknown. We hypothesized that multilevel intracardiac and extracardiac (left femoral vein, coronary sinus, left atrium, pulmonary vein) measurements of several inflammatory proteins (VEGF) would help assessing the extent and the source of inflammation in AF patients.

The measurement of von Willebrand factor (vWF) levels in multiple vascular sites would also help to define the site of endothelial dysfunction and of production of this thrombogenic factor.

Although AF is associated with an increased risk of stroke, the risk is not homogeneous. Permanent and persistent AF are associated with similar thromboembolic risk to that of paroxysmal AF.

ELIGIBILITY:
Inclusion Criteria:

* Patient for which an electrophysiology exploration or ablation is programmed;
* Patient who have given written informed consent.

Exclusion Criteria:

* Pregnant women;
* lung disease history (all sources);
* inflammatory disease history (all types);
* Anti-inflammatory treatment;
* left ventricular ejection fraction <35%;
* history of stroke;
* Participation in other ongoing clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-02; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
VEGF concentration | Day one
  Concentration for VEGF between the peripheral blood and the samples collected from the coronary sinus or the left atrium, as well as a possible difference among patients with paroxysmal AF and those with persistent A. These assays will be carried out by an ELISA technique
vWF concentration | Day one
  Concentration for vWF between the peripheral blood and the samples collected from the coronary sinus or the left atrium, as well as a possible difference among patients with paroxysmal AF and those with persistent A. These assays will be carried out by an ELISA technique

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No